CLINICAL TRIAL: NCT00409864
Title: Endoscopic Versus Percutaneous Biliary Drainage For Hilar Block Due to Carcinoma Gall Bladder: A Randomized Prospective Trial and Quality Of Life Assessment
Brief Title: Endoscopic Versus Percutaneous Drainage For Hilar Block in Gall Bladder Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: VP Gupta, A.I.I.M.S.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIS/1/2003
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2006-12

CONDITIONS: Gallbladder Cancer; Obstructive Jaundice
Keywords: Gallbaldder Cancer; Endoscopic stenting; Percutaneous biliary drainage
MeSH Terms: conditions — Gallbladder Neoplasms; Jaundice, Obstructive

ARMS (2):
- PTBD (Active Comparator): percutaneous biliary drainage
  Interventions: Procedure: Endoscopic biliary stenting, Percutaneous biliary stenting
- Endoscopic stenting (Active Comparator): ERCP and stenting
  Interventions: Procedure: Endoscopic biliary stenting, Percutaneous biliary stenting

INTERVENTIONS:
Procedure: Endoscopic biliary stenting, Percutaneous biliary stenting — percutaneous 10 F stent, endoscopic 10 F stent insertion

SUMMARY:
Cancer of the gallbladder (CaGB) is one of the most common causes of malignant obstructive jaundice. Jaundice is the second most common presentation and occurs in 30-60% of patients with CaGB. It is obstructive in nature and frequently associated with pruritus, which is very disturbing for the patients. The usual mechanism of obstruction is direct infiltration of the bile duct by the tumour. Most patients with CaGB with obstructive jaundice are not amenable to a curative surgical resection and hence effective palliation is the goal of treatment. Although surgical bypass has been the traditional palliative approach, it is associated with substantial morbidity and mortality. Non-operative alternatives in the form of percutaneous and endoscopic drainage are available. A few trials have shown that endoscopic drainage is better than percutaneous drainage in patients with lower end bile duct obstruction due to pancreatic and peri-ampullary cancer. However, the scenario is quite different in patients with upper end of bile duct obstruction as occurs due to CaGB. Endoscopic drainage is associated with a higher incidence of cholangitis in patients with a block at the upper end of the bile duct and the success rate varies from 40% to 80%, while percutaneous drainage may be associated with complications such as biliary leak and bleeding. There has been no randomized trial comparing endoscopic and percutaneous drainage in patients with malignant obstruction due to CaGB. The objective of the present study is to carry out a randomized prospective trial comparing percutaneous and endoscopic biliary drainage in patients with CaGB with obstructive jaundice and to assess their quality of life.

DETAILED DESCRIPTION:
Hypothesis: Percutaneous biliary stenting is superior to endoscopic stenting in providing successful biliary drainage by 20% in patients with unresectable malignant hilar block due to carcinoma of gall bladder.

Background: Malignant biliary obstruction at the liver hilum is caused by a heterogeneous group of tumours that include cholangiocarcinoma, gallbladder cancer (CaGB) and metastatic cancer. CaGB is the commonest cause of malignant hilar obstruction in India (1). Jaundice is the second most common presentation and occurs in 30-60% of patients with CaGB (2-5). It is obstructive in nature and frequently associated with pruritis, which is very disturbing for the patients. Most patients with CaGB with surgical obstructive jaundice are not amenable to a curative surgical resection (5) and hence effective palliation is the goal of treatment. Although surgical bilioenteric bypass has been the traditional palliative approach (6), it is associated with substantial morbidity and mortality. Non-operative alternatives in the form of percutaneous and endoscopic drainage are available (7-8). Unilateral drainage of single liver lobe may be sufficient to palliate the jaundice and, pruritis and improve the quality of life (9-15). A few trials have shown that endoscopic drainage is better than percutaneous drainage in patients with lower end bile duct obstruction due to pancreatic and periampullary cancer. However, the scenario is quite different in patients with hilar malignant obstruction. Endoscopic drainage is associated with a higher incidence of cholangitis in patients with a block at the confluence (Bismuth types 2 and 3) and the success rate varies from 40% to 80%, while percutaneous drainage may be associated with complications such as biliary leak and bleeding. There has been no randomized trial comparing endoscopic and percutaneous drainage in patients with malignant hilar obstruction alone.

Objective: To compare unilateral PTBD and endoscopic stenting in patients with CaGB with hilar block in terms of Successful drainage and Quality of life Patients and Methods Consecutive patients with CaGB and jaundice will be enrolled in the study. The diagnosis of CaGB and biliary obstruction will be established on the basis of an ultrasound of the abdomen and a dual phase CT scan. Histological and/or cytological confirmation of the malignancy will be established wherever possible by doing a FNAC/trucut biopsy. Hilar block will be classified according to the Bismuth Corlette classification based on the preprocedural investigations (16). Final differentiation between type 2 and 3 blocks will be based on findings noted during intervention.

Inclusion criteria CaGB with hilar block not suitable for curative resection with one or more of the following criteria: (i) Jaundice with serum bilirubin >10 mg/dl, (ii) Pruritus, (iii) Cholangitis Exclusion criteria: Poor performance status: Karnofsky index < 60, Type 1 and 4 hilar block, Uncontrolled ascites, Duodenal obstruction, Patients who opted for insertion of a metallic stent.

Sample size calculation: The number of patients to be included was calculated to be 91 patients in each group based on the assumption that percutaneous drainage will be better than endoscopic drainage by 20 %. The sample size was calculated by the formula for a power of 80% and alpha error of 0.05.

The patients will be randomly divided into two groups using random blocks generated by a computer.

Group A - percutaneous biliary drainage (PTBD) Group B - Endoscopic stenting (ES) Pre-procedural preparation(17) Patients will undergo detailed investigations and an informed consent will be obtained.

The procedure will be performed under conscious sedation (midazolam and pentozocine) with a liberal infiltration of local anesthetic at the site and the capsule of the liver for PTBD.

1. PTBD procedure (17) Either a right or left sided approach will be used for PTBD. Once entry will be gained to a suitable duct the standard Seldinger technique will be used to place a guidewire in the biliary system. The tract will be dilated and after crossing the obstruction with a hydrophilic guidewire, a ring biliary catheter will be placed to provide internal-external drainage. In a subsequent session, a 10 F, straight plastic stent (polyurethane) will be placed into the system across the obstruction to provide internal drainage.
2. Endoscopic stenting (18) A therapeutic duodenoscope and a standard sphincterotome will be used for cannulation of the bile duct. A hydrophilic guidewire will be used to cross the malignant stricture. After the stricture is crossed a guide catheter will be passed over the guidewire and then a 10 F straight plastic stent will be inserted across the stricture over the guidewire.

Primary outcome measures:

1. Successful drainage: A decrease in bilirubin to less than 75% of the pretreatment value within 7 days
2. Early cholangitis: Occurring within 48 hours to 7 days of the procedure as evidenced by fever, leukocytosis and worsening LFTs.
3. Quality of life

Secondary outcome measures:

1. Complications
2. Procedure-related and 30-day mortality
3. Stent patency time will be defined by time to stent occlusion.

Hematological and biochemical parameters will be assessed at days 2 and 7, 1 month after stent placement and every 3 months thereafter. Patients will be re-evaluated 7 days, 1 month after stent placement and 3 months thereafter.

Quality of life will be assessed using the WHO-QOL BREF26 and EORTC QLQ-30 questionnaires pre-procedure, at 1 month and at 3 months.

World Health Organization-QOL BREF-26 (19) This has 26 items, which cover physical, psychological, social and environmental domains. The daily activity is graded in accordance with the 5 grade scale of performance status recommended by the WHO. WHO-QOL domain scores will be calculated using the guidelines given in the WHO-QOL scoring manual. A high score represents a high level of QOL.

EORTC QLQ-30 (20) The EORTC QLQ-30 consists of 30 generally applicable items. It incorporates a functional scale (items 1-5), a role functioning scale (item 6,7), a general symptom scale (item 8-19), scales on cognitive (item 20-25), emotional (items 21-24) and social (items 26-27) functioning, financial strain scale (item 28) and global health status scale (item 29,30). Scoring will be done using the EORTC scoring manual.

A high score for a functional scale will represent a high/healthy level of functioning, a high score for global health status/QOL will represent high QOL but a high score for symptom scale/item will represent a higher level of symptomatology/ problem.

All patients will be instructed to contact the department, if any symptom suggestive of a complication appeared. Additional information regarding current status or death will be obtained by direct contact with the referring physician or the patient by telephone/letter.

Statistical analysis Data will be analyzed according to both the intention-to-treat (ITT) and per protocol (PP) methods. The baseline characteristics will be expressed in mean (SD). The Pearson chi -square test and Fischer exact test will be used for comparison of categorical data as appropriate. The t-test will be used for comparison of continuous variables. Cumulative survival will be estimated using Kaplan-Meier life table analysis, and the groups will be compared by log rank chi-square test.

The QOL score analysis will be done using Paired 't' test for comparison between baseline and 1 month and baseline and 3 months within the groups. MANOVA will be used to assess the trend of the scores.

References

1. Malkan G, Mohandas KM. Epidemiology of digestive cancers in India. I. General principles and esophageal cancer. Indian J Gastroenterol 1997;16(3):98-102
2. Wanebo HJ, Castle WN, Fechner RE. Is carcinoma of the gall bladder a curable lesion? Ann Surg 1982;195:624-31.
3. Kelly TR, Chamberlain TR. Carcinoma of the gall bladder. Am J Surg 1982; 143:737-41
4. Morrow CF, Sutherland DE, Florack G, Eisenberg MM, Grage TB. Primary carcinoma gall bladder: Significance of subserosal lesions and results of aggressive surgical treatment and adjuvant chemotherapy. Surgery 1983;94:709-14
5. Kumaran V, Gulati MS, Paul SB, Pande GK, Sahni P, Chattopadhyay TK. The role of dual phase helical CT in assessing respectability of carinoma of the gall bladder. Eur Radiol 2002;12:1993-99.
6. Bismuth H, Castaing D, Traynor O. Resection or palliation; priority of surgery in the treatment of hilar cancer. World J Surg 1988; 12:39-47.
7. Huibregtse K, Tytgat GNJ. Palliative treatment of jaundice by transpapillary introduction of biliary endoprosthesis. Gut 1982; 23:371-5.
8. Cotton PB. Endoscopic methods for relief of malignant obstructive jaundice. World J Surg 1984;8:854-61.
9. Dowsett JF, Vaira D, Hatfield AR, Cairns SR, Polydorou AA, Frost R, et al. Endoscopic biliary therapy using the combined percutaneous and endosopic route. Gastroenterology 1989;96:1180-6.
10. Polydorou AA, Cairns SR, Dowsett JF, Hatfield AR, Salmon PR, Cotton PB, et al. Palliation of proximal malignant biliary obstruction by endoscopic endoprosthesis insertion. Gut 1991;32:685-9.
11. De Palma GD, Galloro G, Sicilliano S, Ivonini P, Catanzano C. Unilateral versus bilateral endoscopic hepatic duct drainage in patients with malignant hilar biliary obstruction: results of a prospective, randomized and controlled study. Gastrointest Endosc 2001;53:547-53
12. Sherman S. Endoscopic drainage of malignant hilar obstruction: is one biliary stent enough or should we place two? Gastrointest Endosc 2001;53:681-4.
13. Chang WH, Kortan P, Haber GB. Outcome in patients with bifurcation tumors who undergo unilateral versus bilateral hepatic duct drainage. Gastrointest Endosc 1998;47:354-62
14. Mehta S, Ozden ZS, Dhanireddy S, Pleskow DP, Chutanni R. Endoscopic single versus double (bilateral) Wallstents for palliation of malignant Bismuth type III/IV hilar strictures: comparison of clinical outcomes and costs (abstract). Gastrointest Endosc 1999;49:AB234.
15. De Palma, Angelo Pezzullo, Maria Rega, Unilateral placement of metallic stents for malignant hilar obstruction: a prospective study. Gastrointest Endosc 2003;55:50-5.
16. Bismuth H, Castaing D, Traynor O. Resection or palliation :priority of surgery in the treatment of hilar cancer. World j Surg 1988;12:39-47.
17. Gulati MS, Srinivasan A, Agarwal PP. Percutaneous Management of Malignant Biliary Obstruction: The Indian Perspective. Tropical Gastroenterology 2003;24:47-58.
18. Ahuja V, Garg PK, Kumar D, Goindi G, Tandon RK. Presence of white bile associated with lower survival in malignant biliary obstruction. Gastrointest Endosc 2002;55:186-91.
19. World Health Organization Handbook for Reporting Results of cancer Treatment. World Health Organization Publication No .48 Geneva World Health Organization 1979.
20. Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst 1993;85:365-76.

ELIGIBILITY:
Inclusion Criteria:

* CaGB with hilar block not suitable for curative resection with one or more of the following criteria:

  * Jaundice with serum bilirubin >10 mg/dl,
  * Pruritus,
  * Cholangitis

Exclusion Criteria:

* Poor performance status: Karnofsky index < 60,
* Type 1 and 4 hilar block,
* Uncontrolled ascites,
* Duodenal obstruction,
* Patients who opted for insertion of a metallic stent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2003-10; Primary Completion 2005-07 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Successful drainage: A decrease in bilirubin to less than 75% of the pretreatment value within 7 days | 7 days
Early cholangitis: Occurring within 48 hours to 7 days of the procedure as evidenced by fever, leukocytosis and worsening LFTs. | 7 days
Quality of life | 30 days

SECONDARY OUTCOMES:
Complications | 30 day
Procedure-related and 30-day mortality | 30 days
Stent patency time will be defined by time to stent occlusion | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Peush Sahni, MS, PhD, Study Director — Dept. of GI Surgery, All India Institute of Medical Sciences, New Delhi, India; Sundeep Saluja, MS, MCh, Principal Investigator — Dept. of GI Surgery, All India Institute of Medical Sciences, New Delhi
Locations (1):
- All India Institute of Medical Sciences,, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Speer AG, Cotton PB, Russell RC, Mason RR, Hatfield AR, Leung JW, MacRae KD, Houghton J, Lennon CA. Randomised trial of endoscopic versus percutaneous stent insertion in malignant obstructive jaundice. Lancet. 1987 Jul 11;2(8550):57-62. doi: 10.1016/s0140-6736(87)92733-4. PMID 2439854
- [Background] Pinol V, Castells A, Bordas JM, Real MI, Llach J, Montana X, Feu F, Navarro S. Percutaneous self-expanding metal stents versus endoscopic polyethylene endoprostheses for treating malignant biliary obstruction: randomized clinical trial. Radiology. 2002 Oct;225(1):27-34. doi: 10.1148/radiol.2243011517. PMID 12354980